CLINICAL TRIAL: NCT02738879
Title: A Phase III, Multicenter, Randomized, Double-Blind, Placebo-Controlled Clinical Trial to Study the Efficacy and Safety of the Continuation of Sitagliptin Compared With the Withdrawal of Sitagliptin During Initiation and Titration of Insulin Glargine (LANTUS®) in Subjects With Type 2 Diabetes Mellitus
Brief Title: Randomized Sitagliptin Withdrawal Study (MK-0431-845)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0431-845; 2015-004990-34 (EudraCT Number); MK-0431-845 (Other: Merck Protocol Number)
Record Dates: First submitted 2016-04-11; First posted 2016-04-14 (Estimated); Results first posted 2019-02-25 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate; Metformin; Insulin Glargine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sitagliptin (Experimental): Sitagliptin 100 mg, oral, once daily for 30 weeks
  Interventions: Drug: Sitagliptin; Drug: Metformin; Drug: Metformin XR; Drug: Insulin glargine
- Placebo (Placebo Comparator): Placebo to sitagliptin, 100 mg, oral, once daily for 30 weeks
  Interventions: Drug: Placebo to sitagliptin; Drug: Metformin; Drug: Metformin XR; Drug: Insulin glargine

INTERVENTIONS:
Drug: Sitagliptin — Sitagliptin 100 mg, oral, once daily for 30 weeks
  Other Names: Januvia®
  Arms: Sitagliptin
Drug: Placebo to sitagliptin — Placebo to sitagliptin, 100 mg, oral, once daily for 30 weeks
  Arms: Placebo
Drug: Metformin — At least 1500 mg/day, oral, twice daily for participants entering the study on immediate-release metformin + sitagliptin or a fixed dose combination (FDC).
Drug: Metformin XR — At least 1500 mg/day, oral, once daily for participants entering the study on extended-release metformin + sitagliptin or a FDC.
Drug: Insulin glargine — Insulin glargine (LANTUS®) initiated at 10 units and titrated based on a treat-to-target algorithm to achieve fasting glucose levels of 72-100 mg/dL (4-5.6 mmol/L); administered once daily subcutaneously.
  Other Names: LANTUS®)

SUMMARY:
This is a trial of continuing sitagliptin versus withdrawing sitagliptin in participants with Type 2 diabetes mellitus (T2DM) and inadequate glycemic control who initiate and titrate insulin glargine (LANTUS®) based on a treat-to-target algorithm to achieve fasting glucose levels of 72-100 mg/dL (4-5.6 mmol/L). A primary hypothesis of this trial is that after 30 weeks, continuing sitagliptin results in a greater reduction of hemoglobin A1C (A1C) relative to withdrawing sitagliptin.

ELIGIBILITY:
Inclusion Criteria:

* Have T2DM based on American Diabetes Association guidelines
* Be on one of the following treatment regimens:

  1. Stable dose of sitagliptin (100 mg/day) and metformin IR or XR (metformin) (≥1500 mg/day) either co-administered or as a fixed dose combination (FDC) for ≥12 weeks with A1C between 7.5% and 11.0%, inclusive.

     OR
  2. Stable dose of metformin (≥1500 mg/day) and another dipeptidyl peptidase-4 (DPP-4) inhibitor (at maximum labeled dose, other than sitagliptin, either co-administered or as a FDC, for ≥12 weeks with A1C between 7.5% and 11.0%, inclusive.

     OR
  3. Stable dose of sitagliptin (100 mg/day) and metformin (≥1500 mg/day) either co administered or as a FDC, and a sulfonylurea for ≥12 weeks OR stable dose of metformin (≥1500 mg/day) and a sulfonylurea administered as a FDC and sitagliptin (100 mg/day) with A1C between 7.0% and 10.0%, inclusive.

     OR
  4. Stable dose of metformin (≥1500 mg/day) and another DPP-4 inhibitor (at maximum labeled dose), other than sitagliptin, either co-administered or as a FDC, and a sulfonylurea for ≥12 weeks OR stable dose of metformin (≥1500 mg/day) and a sulfonylurea administered as a FDC and another DPP-4 inhibitor other than sitagliptin with A1C between 7.0% and 10.0%, inclusive OR
  5. Stable dose of metformin (≥1500 mg/day) and a sulfonylurea either co-administered or as a FDC for ≥12 weeks with A1C between 7.5% and 11.0%, inclusive.
* Meet one of the following categories:

  1. The participant is a male
  2. The participant is a female who is not of reproductive potential
  3. The participant is a female who is of reproductive potential and agrees to avoid becoming pregnant while receiving study drug and for 14 days after the last dose of study drug by practicing abstinence from heterosexual activity OR use (or have her partner use) acceptable contraception during heterosexual activity

Exclusion Criteria:

* Has been treated with any anti-hyperglycemic agent (AHA) other than protocol-specified agents (i.e., other than metformin, DPP-4 inhibitor, or sulfonylurea agent) within the prior 12 weeks.
* Has a history of 2 or more episodes of hypoglycemia resulting in seizure, coma, or loss of consciousness, OR has had recurrent (≥3 times per week) episodes of hypoglycemia over the past 8 weeks.
* Has a history of type 1 diabetes mellitus (T1DM) or ketoacidosis, or has a history of latent autoimmune diabetes of adults (LADA), is assessed by the investigator as possibly having T1DM or LADA confirmed with a C-peptide <0.7 ng/mL (<0.23 nmol/L), or has a history of other specific types of diabetes (e.g., genetic syndromes, secondary pancreatic diabetes, diabetes due to endocrinopathies, drug- or chemical-induced, or post-organ transplant).
* Is assessed by the investigator to be not appropriate for, or does not agree to target, a fasting glucose of 72-100 mg/dL (4.0-5.6 mmol/L).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 746 (Actual)
Dates: Start 2016-05-09 (Actual); Primary Completion 2018-01-22 (Actual); Study Completion 2018-01-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://engagezone.msd.com/doc/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Derived] Roussel R, Duran-Garcia S, Zhang Y, Shah S, Darmiento C, Shankar RR, Golm GT, Lam RLH, O'Neill EA, Gantz I, Kaufman KD, Engel SS. Double-blind, randomized clinical trial comparing the efficacy and safety of continuing or discontinuing the dipeptidyl peptidase-4 inhibitor sitagliptin when initiating insulin glargine therapy in patients with type 2 diabetes: The CompoSIT-I Study. Diabetes Obes Metab. 2019 Apr;21(4):781-790. doi: 10.1111/dom.13574. Epub 2018 Dec 9. PMID 30393950

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 746 participants were randomized across 149 study sites in 22 countries.
Pre-assignment Details: Male and female participants with Type 2 diabetes mellitus (T2DM) ≥18 years of age were enrolled in this trial.
Period: Overall Study
Arm/Group | Sitagliptin | Placebo
Started | 374 | 372
Treated | 373 | 370
Completed | 361 | 347
Not Completed | 13 | 25
Not completed — Adverse Event | 1 | 1
Not completed — Death | 0 | 2
Not completed — Lost to Follow-up | 1 | 5
Not completed — Protocol Violation | 1 | 3
Not completed — Physician Decision | 3 | 4
Not completed — Pregnancy | 0 | 1
Not completed — Screen Failure | 1 | 2
Not completed — Site Discontinued Study Participation | 1 | 0
Not completed — Withdrawal by Subject | 5 | 7

BASELINE CHARACTERISTICS:
Population: The overall number of baseline participants included all randomized participants.
Groups:
- Placebo: Placebo to sitagliptin 100 mg, oral, once daily for 30 weeks
- Total: Total of all reporting groups
Arm/Group | Sitagliptin | Placebo | Total
Number analyzed (Participants) | 374 | 372 | 746
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.5 (9.5) | 58.1 (9.7) | 58.3 (9.6)
Age, Customized [Count of Participants; unit: Participants]
  In utero | 0 | 0 | 0
  Preterm newborn infants (gestational age < 37 wks) | 0 | 0 | 0
  Newborns (0-27 days) | 0 | 0 | 0
  Infants and toddlers (28 days-23 months) | 0 | 0 | 0
  Children (2-11 years) | 0 | 0 | 0
  Adolescents (12-17 years) | 0 | 0 | 0
  Adults (18-64 years) | 275 | 272 | 547
  From 65-84 years | 99 | 100 | 199
  85 years and over | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 204 | 181 | 385
  Male | 170 | 191 | 361
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 19 | 18 | 37
  Asian | 42 | 37 | 79
  Native Hawaiian or Other Pacific Islander | 6 | 1 | 7
  Black or African American | 12 | 12 | 24
  White | 259 | 270 | 529
  More than one race | 34 | 34 | 68
  Unknown or Not Reported | 2 | 0 | 2
Geographic Region [Count of Participants; unit: Participants]
  Asia | 36 | 26 | 62
  Europe | 158 | 172 | 330
  Latin America | 85 | 83 | 168
  North America | 80 | 78 | 158
  Other | 15 | 13 | 28
Hemoglobin A1C (A1C) [Mean (Standard Deviation); unit: Percent A1C] — Percent A1C= Glycated hemoglobin/total hemoglobin x 100 Population: All randomized and treated participants
  Percent A1C
    number analyzed (Participants) | 373 | 370 | 743
    (all) | 8.8 (0.9) | 8.8 (1.0) | 8.8 (0.9)
Fasting Plasma Glucose (FPG) [Mean (Standard Deviation); unit: mg/dL] — Fasting plasma glucose level after a 10-hour overnight fast. Population: All randomized and treated participants
  mg/dL
    number analyzed (Participants) | 373 | 370 | 743
    (all) | 199.0 (50.8) | 201.2 (51.8) | 200.1 (51.3)
Estimated Glomerular Filtration Rate [Mean (Standard Deviation); unit: mL/min/1.73 m^2] — Estimated Glomerular Filtration Rate (eGFR) is a test of renal function. Population: All randomized and treated participants
  mL/min/1.73 m^2
    number analyzed (Participants) | 373 | 370 | 743
    (all) | 103.7 (30.3) | 106.4 (28.1) | 105.1 (29.2)
Body Weight [Mean (Standard Deviation); unit: Kilograms] — Population: All randomized and treated participants
  Kilograms
    number analyzed (Participants) | 373 | 370 | 743
    (all) | 84.8 (19.8) | 85.6 (18.9) | 85.2 (19.4)
Anti-Hyperglycemic Agent [Count of Participants; unit: Participants] — Background Anti-Hyperglycemic Agent (AHA) at Screening metformin = Met) dipeptidyl peptidase 4 inhibitor = DPP-4i
  Participants
    Met + DPP-4i | 184 | 184 | 368
    Met + DPP-4i + sulfonylurea (SU) | 87 | 86 | 173
    Met + SU | 103 | 102 | 205

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in A1C at Week 30
Description: A1C is blood marker used to report average blood glucose levels over prolonged periods of time. Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100. Thus, this change from baseline reflects the Week 30 A1C minus the Week 0 A1C.
Time Frame: Baseline and Week 30
Population: All randomized participants who received at least one dose of study treatment and had at least one measurement of the respective endpoint (baseline or post-baseline).
Measure: Least Squares Mean (95% Confidence Interval); unit: Percent A1C
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 373 | 370
Percent A1C | -1.88 (-1.98) [-1.98 to -1.78] | -1.42 (-1.52) [-1.52 to -1.32]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; A longitudinal data analysis (LDA) model included terms for treatment, AHA treatment at screening (Met + DPP-4i, Met + DPP-4i + SU, Met + SU), time, and the interactions of time by treatment and of time by AHA treatment at screening. Least Squares Means = LSM; Test type: Non-Inferiority — Hypothesis A: After 30 weeks, continuing sitagliptin is non-inferior relative to withdrawing sitagliptin on the change from baseline in A1C. Non-inferiority is declared if the upper bound of the two-sided 95% CI for the difference is less than 0.3%; LDA; Between Group Difference in the LSM = -0.46, 95% CI 2-sided [-0.58 to -0.34]
Statistical Analysis 2: Comparison: Sitagliptin vs Placebo; A LDA model included terms for treatment, AHA treatment at screening (Met + DPP-4i, Met + DPP-4i + SU, Met + SU), time, and the interactions of time by treatment and of time by AHA treatment at screening; Test type: Superiority — Hypothesis B: After 30 weeks, continuing sitagliptin results in a greater reduction of A1C relative to withdrawing sitagliptin; p < 0.001, LDA; Between Group Difference in the LSM = -0.46, 95% CI 2-sided [-0.58 to -0.34]

2. Primary Outcome: Event Rate of Documented Symptomatic Hypoglycemia With Blood Glucose ≤70 mg/dL (≤3.9 mmol/L)
Description: Documented symptomatic hypoglycemia is defined as an event during which typical symptoms of hypoglycemia are accompanied by a measured (e.g., by fingerstick) plasma glucose concentration ≤70 mg/dL (≤3.9 mmol/L). The event rate was the total number of events divided by follow-up time (participant-years), including multiple events from the same participant.
Time Frame: Up to 30 weeks
Population: All randomized participants who received at least one dose of study treatment. Two participants in the sitagliptin group were not included in the primary analysis due to a missing value of a model covariate (race).
Measure: Number (95% Confidence Interval); unit: Events/Participant-Years
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 371 | 370
Events/Participant-Years | 1.55 (1.22) [1.22 to 1.96] | 2.12 (1.70) [1.70 to 2.66]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Calculated via the Negative Binomial Model including terms for treatment, race (i.e., White and Other), region (i.e., Europe, North America, and Other), AHA treatment at screening, baseline A1C value and baseline body weight and an offset for follow-up time (on the natural log scale); Test type: Superiority; p = 0.039, Negative Binomial Model; Event Rate Ratio = 0.73, 95% CI 2-sided [0.54 to 0.98]

3. Primary Outcome: Percentage of Participants Who Discontinued Study Drug Due to an AE
Description: An AE is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to 30 weeks
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 373 | 370
Percentage of participants | 1.3 | 1.6
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Other — 95% CI; Miettinen & Nurminen; Between Group Difference in Percentages = -0.3, 95% CI 2-sided [-2.3 to 1.7]

4. Secondary Outcome: Percentage of Participants With Events of Documented Symptomatic Hypoglycemia With Blood Glucose ≤70 mg/dL (≤3.9 mmol/L)
Description: Documented symptomatic hypoglycemia is defined as an event during which typical symptoms of hypoglycemia are accompanied by a measured (e.g., by fingerstick) plasma glucose concentration ≤70 mg/dL (≤3.9 mmol/L). The incidence (number of participants with ≥1 event divided by number of participants) of documented symptomatic hypoglycemia was determined.
Time Frame: Up to 30 weeks
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 373 | 370
Percentage of participants | 33.5 (28.5) [28.5 to 38.6] | 37.7 (32.7) [32.7 to 42.6]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority; p = 0.250, Miettinen and Nurminen; Between Group Difference in Percentages = -4.1, 95% CI 2-sided [-11.2 to 2.9]

5. Secondary Outcome: Change From Baseline in Total Daily Insulin Dose (Units) at Week 30
Description: Change from baseline reflects the Week 30 total daily insulin dose minus the Week 0 total daily insulin dose. The Week 0 total daily insulin dose was 0, by definition, because insulin was not administered at baseline.
Time Frame: Baseline and Week 30
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: Insulin Units
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 365 | 367
Insulin Units | 53.2 (48.5) [48.5 to 58.0] | 61.3 (56.5) [56.5 to 66.0]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; The analysis is based on a LDA model including terms for treatment, AHA treatment at screening (Met + DPP-4i, Met + DPP-4i + SU, Met + SU), time, and the interactions of time by treatment and of time by AHA treatment at screening; Test type: Superiority; p = 0.016, LDA model; Between Group Difference in the LSM = -8.0, 95% CI 2-sided [-14.6 to -1.5]

6. Secondary Outcome: Event Rate of Documented Hypoglycemia With Blood Glucose ≤70 mg/dL (≤3.9 mmol/L)
Description: Documented hypoglycemia is defined by a measured (e.g., by fingerstick) plasma glucose concentration ≤70 mg/dL (≤3.9 mmol/L). The event rate was the total number of events divided by follow-up time (participant-years), including multiple events from the same participant.
Time Frame: Up to 30 weeks
Population: All randomized participants who received at least one dose of study treatment and had at least one measurement of the respective endpoint (baseline or post-baseline). Two participants (both in the sitagliptin group) were not included in the analysis due to a missing value of a model covariate (race).
Measure: Number (95% Confidence Interval); unit: Events/Participant-Years
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 371 | 370
Events/Participant-Years | 5.05 (4.34) [4.34 to 5.88] | 6.21 (5.33) [5.33 to 7.24]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Negative Binomial Model including terms for treatment, race (i.e., White and Other), region (i.e., Europe, North America, and Other), AHA treatment at screening, baseline A1C value and baseline body weight and an offset for follow-up time (on the natural log scale); Test type: Superiority; p = 0.041, Negative Binomial Model; Event Rate Ratio = 0.81, 95% CI 2-sided [0.67 to 0.99]

7. Secondary Outcome: Event Rate of Documented Hypoglycemia With Blood Glucose <56 mg/dL (≤3.1 mmol/L)
Description: Documented hypoglycemia is defined by a measured (e.g., by fingerstick) plasma glucose concentration <56 mg/dL (≤3.1 mmol/L). The event rate was the total number of events divided by follow-up time (participant-years), including multiple events from the same participant.
Time Frame: Up to 30 weeks
Population: as for outcome 6
Measure: Number (95% Confidence Interval); unit: Events/Participant-Years
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 371 | 370
Events/Participant-Years | 0.30 (0.20) [0.20 to 0.45] | 0.36 (0.25) [0.25 to 0.53]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; [analysis description as in outcome 6, analysis 1]; Test type: Superiority; p = 0.473, Negative Binomial Model; Event Rate Ratio = 0.83, 95% CI 2-sided [0.51 to 1.37]

8. Secondary Outcome: Percentage of Participants With Documented Hypoglycemia With Blood Glucose <56 mg/dL (≤3.1 mmol/L)
Description: Documented hypoglycemia is defined by a measured (e.g., by fingerstick) plasma glucose concentration <56 mg/dL (≤3.1 mmol/L).
Time Frame: Up to 30 weeks
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 373 | 370
Percentage of participants | 12.4 (8.9) [8.9 to 15.8] | 13.6 (10.0) [10.0 to 17.2]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Percentages and difference in percentages were calculated via the Miettinen and Nurminen stratified by AHA treatment at screening. Includes imputed events after participants discontinued from the study medication, using a Gamma frailty model. The bootstrap method was used to obtain the CI and p-value; Test type: Superiority; p = 0.624, Miettinen and Nurminen; Between Group Difference in Percentages = -1.2, 95% CI 2-sided [-6.2 to 3.7]

9. Secondary Outcome: Percentage of Participants With A1C Goal <7.0% (<53 mmol/Mol) at Week 30
Description: A1C is blood marker used to report average blood glucose levels over prolonged periods of time. Percentage A1C is the ratio of glycated hemoglobin to total hemoglobin x 100.
Time Frame: Week 30
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 373 | 370
Percentage of participants | 54.2 | 35.4
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority; p < 0.001, Miettinen and Nurminen; Between Group Difference in Percentages = 18.8, 95% CI 2-sided [11.6 to 25.7]

10. Secondary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Week 30
Description: Blood glucose was measured on a fasting basis. Blood was drawn at predose on Day 1 and after 30 weeks of treatment to determine change in plasma glucose levels (i.e., FPG at Week 30 minus FPG at Week 0).
Time Frame: Baseline and Week 30
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: mg/dL
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 373 | 370
mg/dL | -84.8 (-90.0) [-90.0 to -79.6] | -78.3 (-83.5) [-83.5 to -73.1]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Analysis was based on a LDA model including terms for treatment, AHA treatment at screening (Met + DPP-4i, Met + DPP-4i + SU, Met + SU), time, and the interactions of time by treatment and of time by AHA treatment at screening; Test type: Superiority; p = 0.020, LDA; Between Group Difference in the LSM = -6.5, 95% CI 2-sided [-11.9 to -1.0]

11. Primary Outcome: Percentage of Participants Who Experienced One or More Adverse Events (AEs)
Description: as for outcome 3
Time Frame: Up to 32 weeks
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 373 | 370
Percentage of participants | 57.9 | 60.0
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Other — 95% CI; Miettinen & Nurminen; Between Group Difference in Percentages = -2.1, 95% CI 2-sided [-9.1 to 5.0]

12. Secondary Outcome: Event Rate of Documented Symptomatic Hypoglycemia With Blood Glucose <56 mg/dL (≤3.1 mmol/L)
Description: Documented symptomatic hypoglycemia is defined as an event during which typical symptoms of hypoglycemia are accompanied by a measured (e.g., by fingerstick) plasma glucose concentration <56 mg/dL (≤3.1 mmol/L). The event rate was the total number of events divided by follow-up time (participant-years), including multiple events from the same participant.
Time Frame: Up to 30 weeks
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: Events/Participant-Years
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 371 | 370
Events/Participant-Years | 0.17 (0.10) [0.10 to 0.28] | 0.22 (0.14) [0.14 to 0.36]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; The analysis was calculated via the Negative Binomial Model including terms for treatment, race (i.e., White and Other), region (i.e., Europe, North America, and Other), AHA treatment at screening, baseline A1C value and baseline body weight and an offset for follow-up time (on the natural log scale); Test type: Superiority; p = 0.394, Negative Binomial Model; Event Rate Ratio = 0.76, 95% CI 2-sided [0.40 to 1.44]

13. Secondary Outcome: Percentage of Participants With Documented Hypoglycemia With Blood Glucose ≤70 mg/dL (≤3.9 mmol/L)
Description: Documented hypoglycemia is defined by a measured (e.g., by fingerstick) plasma glucose concentration ≤70 mg/dL (≤3.9 mmol/L).
Time Frame: Up to 30 weeks
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 373 | 370
Percentage of participants | 66.8 (61.9) [61.9 to 71.7] | 68.0 (63.2) [63.2 to 72.9]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; The analysis included imputed events after participants discontinued from the study medication, using a Gamma frailty model. Proportions and difference in proportions were calculated via the Miettinen and Nurminen stratified by AHA treatment at screening. The bootstrap method was used to obtain the CI and p-value; Test type: Superiority; p = 0.740, Miettinen and Nurminen; Between Group Difference in Percentages = -1.2, 95% CI 2-sided [-8.2 to 5.8]

14. Secondary Outcome: Percentage of Participants With Documented Symptomatic Hypoglycemia With Blood Glucose <56 mg/dL (≤3.1 mmol/L)
Description: Documented symptomatic hypoglycemia is defined as an event during which typical symptoms of hypoglycemia are accompanied by a measured (e.g., by fingerstick) plasma glucose concentration <56 mg/dL (≤3.1 mmol/L).
Time Frame: Up to 30 weeks
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 373 | 370
Percentage of participants | 7.6 (4.9) [4.9 to 10.3] | 8.3 (5.4) [5.4 to 11.2]
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Percentages and difference in percentages were calculated via the Miettinen and Nurminen stratified by AHA treatment at screening. The analysis included imputed events after subjects discontinued from the study medication, using a Gamma frailty model. The bootstrap method was used to obtain the CI and p-value; Test type: Superiority; p = 0.712, Miettinen and Nurminen; Between Group Difference in Percentages = -0.7, 95% CI 2-sided [-4.7 to 3.2]

15. Secondary Outcome: Percentage of Participants With A1C Goal <7.0% (<53 mmol/Mol at Week 30 and No Documented Hypoglycemia With Blood Glucose ≤70 mg/dL (≤3.9 mmol/L) up to Week 30
Description: as for outcome 9
Time Frame: Week 30
Population: All randomized participants who received at least one dose of study treatment.
Measure: Number; unit: Percentage of participants
Arm/Group | Sitagliptin | Placebo
Number analyzed (Participants) | 373 | 370
Percentage of participants | 15.3 | 10.0
Statistical Analysis 1: Comparison: Sitagliptin vs Placebo; Test type: Superiority; p = 0.030, Miettinen and Nurminen; Between Group Difference in Percentages = 5.3, 95% CI 2-sided [0.5 to 10.1]

ADVERSE EVENTS:
Time Frame: Up to 32 weeks
Description: The analysis population consisted all randomized participants who received at least one dose of study treatment. Events of hypoglycemia of any type were collected as efficacy endpoints in this study. AEs of symptomatic hypoglycemia could also be reported by investigators.
Arm/Group | Sitagliptin | Placebo
All-Cause Mortality (participants affected / at risk) | 0/373 | 2/370
Serious Adverse Events (participants affected / at risk) | 14/373 | 18/370
Other Adverse Events (participants affected / at risk) | 79/373 | 72/370
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=373) | Placebo (N=370)
Acute myocardial infarction (Cardiac disorders) | 1 (1) | 1 (1)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 0 (0)
Coronary artery disease (Cardiac disorders) | 1 (1) | 1 (1)
Myocardial infarction (Cardiac disorders) | 0 (0) | 1 (1)
Phimosis (Congenital, familial and genetic disorders) | 0 (0) | 1 (1)
Colitis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Strangulated umbilical hernia (Gastrointestinal disorders) | 1 (1) | 0 (0)
Cholecystitis acute (Hepatobiliary disorders) | 1 (1) | 0 (0)
Bronchitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 1 (1) | 0 (0)
Groin abscess (Infections and infestations) | 1 (1) | 0 (0)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
Sialoadenitis (Infections and infestations) | 1 (1) | 0 (0)
Tracheitis (Infections and infestations) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Fibula fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Heart rate irregular (Investigations) | 0 (0) | 1 (1)
Hyponatraemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Endometrial adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Gastrointestinal tract adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Non-Hodgkin's lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1)
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Carotid artery stenosis (Nervous system disorders) | 0 (0) | 1 (1)
Cerebral ischaemia (Nervous system disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 2 (2)
Ischaemic stroke (Nervous system disorders) | 0 (0) | 2 (2)
Lumbar radiculopathy (Nervous system disorders) | 0 (0) | 1 (1)
Neuralgia (Nervous system disorders) | 0 (0) | 1 (1)
Sciatica (Nervous system disorders) | 1 (1) | 0 (0)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0)
Diabetic foot (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin (N=373) | Placebo (N=370)
Nasopharyngitis (Infections and infestations) | 24 (30) | 32 (35)
Hypoglycaemia (Metabolism and nutrition disorders) | 35 (96) | 24 (74)
Headache (Nervous system disorders) | 25 (36) | 19 (23)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results. Sponsor review can be expedited to meet publication timelines.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-07-14): https://cdn.clinicaltrials.gov/large-docs/79/NCT02738879/Prot_SAP_000.pdf